CLINICAL TRIAL: NCT03897218
Title: Dietary Modulation of Intestinal Microbiota as Trigger of Liver Health: Role of Bile Acids - "A Diet for Liver Health (ADLH)"
Brief Title: Dietary Modulation of Intestinal Microbiota as Trigger of Liver Health: Role of Bile Acids - "A Diet for Liver Health"
Acronym: ADLH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-105
Record Dates: First submitted 2019-03-14; First posted 2019-04-01 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Liver health; Diet; Microbiom
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Placebo Comparator): Patients consuming placebo (millet flakes) each day
  Interventions: Dietary Supplement: millet flakes
- Group 2 (Experimental): Patients consuming oatmeal flakes with a low dosage of prebiotic food supplements
  Interventions: Dietary Supplement: oatmeal flakes with prebiotic food supplements
- Group 3 (Experimental): Patients consuming oatmeal flakes with a high dosage of prebiotic food supplements
  Interventions: Dietary Supplement: oatmeal flakes with prebiotic food supplements

INTERVENTIONS:
Dietary Supplement: oatmeal flakes with prebiotic food supplements — The study participants should consume the prescribed amount of the study product every day. The intake should be divided into 1-2 meals. It is not necessary to limit or change normal eating habits.
  Arms: Group 2; Group 3
Dietary Supplement: millet flakes — The study participants should consume the prescribed amount of the study product every day. The intake should be divided into 1-2 meals. It is not necessary to limit or change normal eating habits.
  Arms: Group 1

SUMMARY:
Studies in recent years have demonstrated that the commensal intestinal flora (microbiome) plays a key role in the development of nonalcoholic steatohepatitis (NASH). An unfavourable microbiom can trigger disease development and progression. On the other hand, recent data show that modulation of the microbiom by a diet can prevent the developement of a NASH. Mechanisms of interaction between nutrition, microbiome, intestine and liver are largely unknown. In this research project, the effect of a fibre-rich oat bran on NASH will therefore be investigated. A better understanding of the interaction between diet, microbiome, intestine and liver could form the basis for new preventive therapies of NASH.

DETAILED DESCRIPTION:
In recent years, the results of animal experiments and some human intervention studies indicate that the commensal intestinal flora (microbiome) plays a key role in the development of nonalcoholic steatohepatitis (NASH). An unfavourable composition of the microbiome can trigger disease development and progression. On the other hand, recent data show that modulation of the microbiome through diet, such as a high-fibre diet, can prevent the developement of a NASH. It has been shown that the uptake of fibre-rich oats reduces LDL and total cholesterol without altering the HDL cholesterol level. Indeed, the results of several human intervention studies suggest that a regular intake of oat flakes with prebiotic food supplements is sufficient to lower LDL and total cholesterol levels. In a small clinical trial it was also shown that an intake of oat bran with prebiotic food supplements in two servings per day was associated with a significant reduction in ALT and AST activity in the serum of overweight individuals with signs of altered liver function. In addition, the use of oat bran to influence postprandial glucose and insulin response and satiety was discussed.

However, the mechanisms underlying the positive effects of treatments with pro-, pre- or synbiotics are not yet fully understood and generally accepted therapeutic strategies are still lacking. The exact influence of a fibre-rich diet on intestinal microbiom and bile acid composition is not yet known. In the research project described, the effect of oat bran with prebiotic food supplements on NASH will be investigated and mechanisms of interaction between diet, microbiome, bile acids and liver will be uncovered. A better understanding of this interaction could form the basis for new preventive therapies of NASH.

ELIGIBILITY:
Inclusion Criteria:

* Fatty liver disease diagnosed by sonography (steatosis hepatis grade II and III) and CAP measurement (> 280dB)
* compliance

Exclusion Criteria:

* Allergy to oats
* Alcohol intake of more than 30 g/d (men) or 20 g/d (women)
* Treatment with ursodeoxycholic acid (UDCA), vitamin E or other NASH drugs 3 months prior to randomization
* Hepatocellular carcinoma or non-hepatic malignancy within the last 5 years
* Evidence of cirrhosis of the liver (Child A, B, C) or a history of decompensation
* Liver diseases not related to NASH, including chronic viral hepatitis B/D or C, autoimmune hepatitis, Wilson's disease or clinically manifest iron overload (heterozygous HFE is permitted), cholestatic liver disease (PBC/PSC)
* Adiposity surgery in the last 5 years
* BMI <18.5 kg / m2
* Liver transplantation
* Fibroscan> 12 kPa (patients with liver cirrhosis)
* Lack of CAP and ultrasound evaluation
* Age > 75 years
* HIV infection
* Heart Failure (New York Heart Association Class III - IV)
* Myocardial infarction, unstable coronary artery disease, coronary artery intervention or stroke in the last 6 months
* Unstable COPD, chronic inflammatory bowel disease or rheumatoid arthritis
* Unstable renal failure (changes in serum creatinine > 50% in the last 3 months) or terminal renal failure requiring dialysis
* Uncontrolled hypertension (SBP / DBP> 180/90 despite therapy)
* Uncontrolled metabolic conditions (poorly controlled or decompensated diabetes mellitus, HbA1c >7.5%)
* Food allergies or intolerances that require strict adherence to a diet, such as lactose intolerance or celiac disease.
* Pregnancy or breastfeeding women (anamnesis)
* Treatment with drugs or substances that can induce secondary NASH (e.g., tamoxifen, corticosteroids, amiodarone, methotrexate) or alleviate NASH (TNF antagonists) (e.g. metformin)
* Use of herbal food supplements
* Any participant who has taken antibiotics 6 weeks prior to the study

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the influence of a dietary supplement in oat bran on the course of disease in the early stages of NASH by CAP (Controlled Attenuation Parameter) measurement to determine liver steatosis. | 20 weeks
  CAP measurement (dB/m)
Evaluation of the influence of a dietary supplement in oat bran on the course of disease in the early stages of NASH by determination ALT-concentration in blood samples. | 20 weeks
  Determination of ALT concentration (U/l) in blood samples

SECONDARY OUTCOMES:
Influence of dietary supplement in oat bran on concentration of AST | 20 weeks
  Determination of AST concentration (U/l) in blood samples
Influence of dietary supplement in oat bran on the concentration of gamma-GT | 20 weeks
  Determination of gamma-GT concentration (U/l) in blood samples
Influence of dietary supplement in oat bran on liver steatosis | 20 weeks
  Sonography - Performing an abdominal ultrasound examination to detect liver steatosis
Influence of dietary supplement in oat bran on bile acid metabolism | 20 weeks
  Determination of bile acid composition in stool samples
Influence of dietary supplement in oat bran on the composition of the intestinal microbiome | 20 weeks
  Determination of microbiom in stool samples (bacterial DNA and RNA are isolated from the stool to determine the microbial composition)
Influence of dietary supplement in oat bran on intestinal permeability marker like citrullin | 20 weeks
  Determination of intestinal permeability marker like citrullin (µmol/l)
Influence of dietary supplement in oat bran on metabolic markers | 20 weeks
  Determination of concentration of diffenrent, previously not defined metabolic markers in blood samples by untargeted metabolomics analysis
Influence of dietary supplement in oat bran on inflammatory markers of NASH | 20 weeks
  Determination of concentration of previously not defined inflammatory markers of NASH in blood samples by multiplex assays
Influence of dietary supplement in oat bran on blood pressure | 20 weeks
  Measurement of blood pressure (mmHg)
Assessment of quality of life | 20 weeks
  Questionnaires to evaluate quality of life: EQ-5D-5L EQ-5D questionnaires with 5-point Likert scale: "having no problems", "having slight problems", "having moderate problems", "having severe problems" & "being unable to do/having extreme problems" (the answers euquals 1-5 points, with 5 points beeing the worst outcome)
Assessment of the feeling of satiety/gastrointestinal symptoms | 20 weeks
  Questionnaire "Structured Assessment of Gastrointestinal Symptoms" (SAGIS):
  5-point Likert scale from no problem, mild, moderate, severe and very severe problem (0-4 points; 4 points equals "very severe problem"

CONTACTS AND LOCATIONS:
Overall Officials: Christian Trautwein, Prof. Dr., Principal Investigator — Uniklinik RWTH Aachen, Med. Klinik III
Locations (3):
- Medical University of Vienna, Vienna, Austria
- University Hospital RWTH Aachen, Aachen, Germany
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Brandt A, Yergaliyev T, Halibasic E, Cyba A, Jaeger JW, Gong R, Hernandez-Arriaga A, Schneider CV, Sjoland W, Molinaro A, Trauner M, Trautwein C, Camarinha-Silva A, Bergheim I, Schneider KM. Fiber enrichment is not superior to dietary monitoring in MASLD: A dual-center, double-blind, placebo-controlled trial. iScience. 2025 Nov 11;28(12):114019. doi: 10.1016/j.isci.2025.114019. eCollection 2025 Dec 19. PMID 41438070